CLINICAL TRIAL: NCT05908357
Title: Effects of Exergaming on Gait and Fall Risk in Children With Autism Spectrum Disorder (ASD): A Randomized Controlled Clinical Trial
Brief Title: Study of Two Exercises Protocols for Autism Spectrum Disorder
Acronym: STEP-TEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, KAREN VALADARES TRIPPO, Professor, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 66594723.2.0000.5543
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: AUTISM SPECTRUM DISORDER; GAIT; ACIDENTAL FALLS; EXERGAMING; PHYSICAL THERAPY MODALITIES
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both assessors participating in the study will be masking for the group of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming Group (EG) (Experimental): The EG will participate in the intervention protocol with exergaming and will also receive the guidance booklet at the end of the treatment. Protocol: twice a week, with a total duration of 40-45 minutes each, conducted by a single physiotherapist. The initial 10 minutes will be for reception, accommodation/heating and anticipation of the service. The Exergaming will last 25-30 minutes, observing the children's reactions to the dosage of the game and the manual and verbal interventions of the physiotherapist. The final 5 minutes will be for cooling down (relaxing music).
  The video game will be the Xbox 360 with a Kinect TM sensor , which captures body movement during the game. The game will be "Kinect Adventures!", and minigames: "peak of reflections" and "20,000 leaks". During the game, the physiotherapist will stimulate the child's proprioception in order to promote sensory and verbal feedback. The intervention will last 12 weeks, with 2 weekly sessions, totaling 24 sessions.
  Interventions: Other: Exergaming
- Control Group (CG) (Active Comparator): The CG will be formed by participants admitted to the institution and who are on the waiting list for physiotherapy care and will follow the guidelines of the physiotherapy booklet with recommendations for physical activities that encourage the child's usual mobility, such as: moments of play with the family, walks outdoors and encourage varied ludic motor experiences. This booklet will be created by the researcher and will not change the routine of the service. The CG will be telemonitored biweekly via messaging application by the researcher, through a personal telephone, with a proposal to check the progress of the application of the booklet, clarify doubts with the family and monitor the child. This telemonitoring protocol was established exclusively for the research.
  Interventions: Other: Booklet

INTERVENTIONS:
Other: Exergaming — Use of the exergame XboX 360 series with kinect sensor
  Arms: Exergaming Group (EG)
Other: Booklet — Use of the booklet with instructions of exercises to be done at home with tele-health through whatsapp app.
  Arms: Control Group (CG)

SUMMARY:
Introduction: Autism Spectrum Disorder (ASD) is characterized as a neurodevelopmental disorder, with motor symptoms that may predispose to falls and gait changes. Exercises through virtual reality (exergaming) showed good results in children with ASD, but no studies were found that evaluated the effects of exergaming on gait and the risk of falls. Objective: To evaluate the effects of exergaming on motor performance during gait and the risk of falls in children with ASD. Method: Pilot study of a clinical trial. There will be 22 participants, diagnosed with ASD, level I or II; age: 5 to 9 years old; that they do not use medications that interfere with postural balance and falls; without physiotherapy care for at least 2 months. They will be divided into Exergaming Group (EG, n=11) and Control Group (GC, n=11). The GC will receive guidance through booklets. The EG will be submitted to a treatment with exergaming for 3 months, with 2 weekly sessions of 45 min each (initial 10 min, 25-30 of exergaming with the Xbox360 console with Kinect sensor and game "Kinect Adventures!", 5 min of cool down ). They will be assessed using CARS-BR (Childhood Autism Rating Scale - Brazilian version), DCDQ (Developmental Coordination Disorder Questionnaire), EEP (Pediatric Equilibrium Scale), a semi-structured questionnaire to assess the history of falls and prevalence of falls, an adapted motivational scale for ASD, a satisfaction survey, and three-dimensional assessment of gait through the Gait Laboratory. Descriptive analysis will be performed and continuous variables will be summarized in mean and standard deviation, and categorical variables in absolute and relative frequencies. To compare the independent and paired variables, parametric tests will be used and a significance level of 5% will be considered (p <0.05). Pearson's correlation will be used to assess correlations between continuous variables and the Chi square test to assess the relationship between categorical variables. Expected results: It is expected that children from the EG will obtain better results than the CG on gait variables and the risk of falling, with clinical and statistical significance.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder with altered motor aspects, present among 50-88% of children with ASD1. They can present difficulties in motor planning, altered gait, postural imbalance, and decreasing postural control, thus increasing the risk of falls.

Children with ASD have variability in gait patterns intra-individually, considering stride length, stride time, and walking speed5. The gait kinematic alteration includes wider step width, decrease in gait velocity, increase in stance time, gait cycle and step time, and differences in cadence and gait cycle compared to children without ASD5. A study showed that children with ASD have a more severely impaired postural balance than other neurodevelopmental disorders and typical children.

The impaired gait patterns can lead to pain, fatigue, and joint stress, affecting the functional capacity of children with ASD and impacting their quality of life. Also, it has been suggested that the motor alterations present in children with ASD are related to difficulties in communication and socialization, difficulties in the development of cognitive abilities, contribute to adaptative dysfunction, decrease the physical functional capacity, and increase the chance of obesity. The motor abilities are strongly related to adaptative function and quality of life of children with ASD, anticipating the deficits in social communication.

Although there is evidence in the literature concerning motor difficulties in children with ASD, it is estimated that 1,34% of them are diagnosed with motor alteration. Besides, it is an underestimated diagnostic among physical therapists in clinical practice. This highlights the importance of functional diagnostics and the study of possible interventions that can be useful in clinical practice in treating motor alterations, especially gait, and the risk of falls.

Exergaming (EXG) has been used as a treatment in children with ASD, demonstrating positive results. Among the effects of EXG in children with ASD are an improvement in explosive strength, better performance in velocity and agility, improvement of aerobic capacity, better work memory capacity, better strength and agility, improved perception of competence, reduced stereotypical behaviors, improved measurement of executive function, reduced aimless arm movements, and decreased body mass index.

Thus, EXG is a valuable tool to treat children with ASD. However, few studies have used EXG to treat motor aspects, especially those related to gait or balance performance. This highlights the following question: Could EXG improve the gait and lessen the risk of falls in children with ASD? Therefore, the primary objective of this study is to describe a randomized and controlled clinical trial protocol to verify the effect of EXG on gait and risk of falls in children with ASD. The secondary objective is to describe the gait measurement and the risk of falls to assess the effect of exergaming in children with ASD. The hypothesis is that the EXG will lessen gait alterations in children with ASD and improve postural balance, lessening the risk of falls.

ELIGIBILITY:
Inclusion Criteria:

* Children with ASD levels I or II;
* Age 5 to 9 years
* No use of medications that interfere with balance and falls;
* Who have not been undergoing physiotherapeutic care in the last 2 months
* Who present some gait alteration.

Exclusion Criteria:

* Children with genetic syndromes duly diagnosed in association with ASD, based on the medical report;
* Physical disability, respiratory disease, or cardiac complications that prevent exercise;
* Proven hearing or visual loss without the use of hearing aids or eyeglasses respectively;
* With a history of epilepsy/seizures in the last six months and without the use of specific medication;
* Children who, even with the formal consent of those responsible for them, do not accept to participate in the research.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change in performance of gait evaluated through gait analysis - stride length, cadence, velocity, distribution of standing support, size of the support base, oscillation of the center of balance during walking | pre-intervention and immediately after the intervention
  Gait analysis in the tridimensional laboratory of gait
Change in the risk of falls evaluated through Pediatric Balance Scale [description above] | pre-intervention and immediately after the intervention
  Cutoff point for predicting falls is 36 points for children

SECONDARY OUTCOMES:
Prevalence of falls evaluated through a questionnaire about falls [description above] | pre-intervention and immediately after the intervention
  Number and frequency of falls, when the child falls most frequently and the circumstance of the last fall
Changes in postural balance evaluated through Pediatric Balance Scale [description above] | pre-intervention and immediately after the intervention
  Maximum of 56 points, which means ability to perform all tasks
Changes in coordination evaluated through DCDQ [description above] | pre-intervention and immediately after the intervention
  For a 5 year-old-child: from 15 to 46 means problem in coordination; For a 8 year-old-child to 9 year-old-child: from 15 to 55 means problem in coordination
Changes in the motivation about exercising evaluated through an adapted motivational scale for ASD [description above] | pre-intervention and immediately after the intervention
  0 means not motivated; 1-3 less motivation; 4-7 moderated motivation; 8-10 great motivation
Level of Satisfaction through questionnaire [description above] | pre-intervention and immediately after the intervention
  0 means dissatisfaction; 1-3 less satisfaction; 4-7 moderated satisfaction; and 8-10 means great satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Milena V Deitos, Msc Student, Study Chair — Federal University of Bahia
Locations (1):
- Instituto Baiano de Reabilitação - Fundação José Silveira, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson-Hanley C, Tureck K, Schneiderman RL. Autism and exergaming: effects on repetitive behaviors and cognition. Psychol Res Behav Manag. 2011;4:129-37. doi: 10.2147/PRBM.S24016. Epub 2011 Sep 16. PMID 22114543
- [Background] Lim YH, Partridge K, Girdler S, Morris SL. Standing Postural Control in Individuals with Autism Spectrum Disorder: Systematic Review and Meta-analysis. J Autism Dev Disord. 2017 Jul;47(7):2238-2253. doi: 10.1007/s10803-017-3144-y. PMID 28508177
- [Background] Fang Q, Aiken CA, Fang C, Pan Z. Effects of Exergaming on Physical and Cognitive Functions in Individuals with Autism Spectrum Disorder: A Systematic Review. Games Health J. 2019 Apr;8(2):74-84. doi: 10.1089/g4h.2018.0032. Epub 2018 Oct 17. PMID 30332294
- [Background] Lamb SE, Jorstad-Stein EC, Hauer K, Becker C; Prevention of Falls Network Europe and Outcomes Consensus Group. Development of a common outcome data set for fall injury prevention trials: the Prevention of Falls Network Europe consensus. J Am Geriatr Soc. 2005 Sep;53(9):1618-22. doi: 10.1111/j.1532-5415.2005.53455.x. PMID 16137297
- [Background] Rafiei Milajerdi H, Sheikh M, Najafabadi MG, Saghaei B, Naghdi N, Dewey D. The Effects of Physical Activity and Exergaming on Motor Skills and Executive Functions in Children with Autism Spectrum Disorder. Games Health J. 2021 Feb;10(1):33-42. doi: 10.1089/g4h.2019.0180. Epub 2020 Dec 23. PMID 33370161
- [Background] Ries LG, Michaelsen SM, Soares PS, Monteiro VC, Allegretti KM. Cross-cultural adaptation and reliability analysis of the Brazilian version of Pediatric Balance Scale (PBS). Rev Bras Fisioter. 2012 Jun;16(3):205-15. doi: 10.1590/s1413-35552012005000026. Epub 2012 Jun 14. English, Portuguese. PMID 22699691
- [Background] Toscano CVA, Carvalho HM, Ferreira JP. Exercise Effects for Children With Autism Spectrum Disorder: Metabolic Health, Autistic Traits, and Quality of Life. Percept Mot Skills. 2018 Feb;125(1):126-146. doi: 10.1177/0031512517743823. Epub 2017 Dec 9. PMID 29226773
- [Background] Wu YT, Tsao CH, Huang HC, Yang TA, Li YJ. Relationship Between Motor Skills and Language Abilities in Children With Autism Spectrum Disorder. Phys Ther. 2021 May 4;101(5):pzab033. doi: 10.1093/ptj/pzab033. PMID 33522583
- [Background] Zampella CJ, Wang LAL, Haley M, Hutchinson AG, de Marchena A. Motor Skill Differences in Autism Spectrum Disorder: a Clinically Focused Review. Curr Psychiatry Rep. 2021 Aug 13;23(10):64. doi: 10.1007/s11920-021-01280-6. PMID 34387753